CLINICAL TRIAL: NCT00047242
Title: The Pharmacokinetic and Safety Profile of UCN-01 in Combination With Irinotecan in Solid Tumors (Primarily Lung, Ovarian and GI Cancers)
Brief Title: UCN-01 and Irinotecan in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: JHOC-J0173, CDR0000257566; U01CA070095 (NIH); P30CA006973 (NIH); JHOC-J0173; NCI-5528
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2010-08-09 (Estimated); Status verified 2010-08

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — 7-hydroxystaurosporine; Irinotecan

INTERVENTIONS:
Drug: 7-hydroxystaurosporine
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: UCN-01 may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining UCN-01 with chemotherapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining UCN-01 with irinotecan in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and recommended phase II dose of UCN-01 and irinotecan in patients with advanced solid tumors, primarily lung, ovarian, and gastrointestinal tumors.
* Determine the acute and chronic toxicity profile of this regimen in these patients.
* Determine the pharmacokinetics of this regimen in these patients.
* Determine, preliminarily, the anti-tumor effect of this regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive UCN-01 IV over 3 hours on day 1 and irinotecan IV over 90 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of UCN-01 and irinotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the recommended phase II dose.

Patients are followed at 1 month.

PROJECTED ACCRUAL: Approximately 20-30 patients will be accrued for this study within 7-15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative therapy does not exist or is no longer effective

  * Gastrointestinal, lung, and ovarian malignancies are given priority
* No brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 3 months

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin normal
* AST/ALT no greater than 2.5 times upper limit of normal (ULN)

Renal

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular

* No symptomatic coronary artery disease
* No symptomatic cardiac dysfunction
* No symptoms suggestive of coronary artery disease
* LVEF at least 50%

Pulmonary

* No symptomatic pulmonary dysfunction
* FEV_1 greater than 75% of predicted
* DLCO greater than 75% of predicted

Other

* Amylase no greater than 2 times ULN
* No other concurrent uncontrolled illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No diabetes mellitus or random glucose more than 200 mg/dL
* No prior allergic reaction attributed to compounds of similar biological or chemical composition to UCN-01 or irinotecan (including rash and systemic allergic reaction causing hypotension and respiratory distress)
* No chronic diarrhea (more than 5 stools/day)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for 14 days before, during, and for at least 30 days after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* Prior UCN-01 and irinotecan allowed

Endocrine therapy

* Not specified

Radiotherapy

* At least 4 weeks since prior radiotherapy and recovered
* No prior mediastinal radiation

Surgery

* Not specified

Other

* At least 14 days since prior warfarin
* No concurrent warfarin unless required for maintaining patency of existing, permanent IV catheters
* No concurrent commercial or other investigational anticancer agents or therapies
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2002-08; Primary Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ross C. Donehower, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Result] Jimeno A, Rudek MA, Purcell T, Laheru DA, Messersmith WA, Dancey J, Carducci MA, Baker SD, Hidalgo M, Donehower RC. Phase I and pharmacokinetic study of UCN-01 in combination with irinotecan in patients with solid tumors. Cancer Chemother Pharmacol. 2008 Mar;61(3):423-33. doi: 10.1007/s00280-007-0485-9. Epub 2007 Apr 12. PMID 17429623